CLINICAL TRIAL: NCT02312310
Title: Dietary Cocoa Flavanols and Age-Related Memory Decline
Brief Title: Dietary Flavanols and Dentate Gyrus Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Mars, Inc. (Industry)
Responsible Party: Principal Investigator, Richard Sloan, Research Scientist / Professor of Behavioral Medicine (in Psychiatry), New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 7034
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Memory Loss
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- F 0 mg (Placebo Comparator): daily consumption of capsules containing 0 mg cocoa flavanol for 12 weeks
  Interventions: Dietary Supplement: Cocoa Flavanol
- F 260 mg (Active Comparator): daily consumption of capsules containing 260 mg* cocoa flavanol for 12 weeks
  *see note in Record Log regarding the change in the method of assessment of cocoa flavanol content of the capsules
  Interventions: Dietary Supplement: Cocoa Flavanol
- F 510 mg (Active Comparator): daily consumption of capsules containing 510 mg cocoa flavanol for 12 weeks
  Interventions: Dietary Supplement: Cocoa Flavanol
- F 770 mg (Active Comparator): daily consumption of capsules containing 770 mg cocoa flavanol for 12 weeks
  Interventions: Dietary Supplement: Cocoa Flavanol

INTERVENTIONS:
Dietary Supplement: Cocoa Flavanol — 12 weeks administration of cocoa flavanol

SUMMARY:
to assess the effect of differing amounts of a cocoa-derived dietary flavanol (epicatechin ) on dentate gyrus function and corresponding cognitive function

DETAILED DESCRIPTION:
In this double blinded trial, the participants, age 50-75 years, will be randomized to receive 0, 260, 510, or 770 mg daily* for 12 weeks and will be tested before and after the intervention. Cognitive testing will be conducted prior to randomization, and at weeks 4, 12, and 20 of the study.

In an optional substudy, fMRI (functional magnetic resonance imaging) with gadolinium contrast will be conducted to measure dentate gyrus function before randomization and then after completion of the 12-week intervention portion of the trial.

*see note in Record Log regarding the change in the method of assessment of cocoa flavanol content of the capsules

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject). Telephone Screen

  2. Healthy Male or Female subjects. (Females must be post-menopausal) Telephone Screen

  3. Age between 50 and 75 years, both inclusive. Telephone Screen

  4. Body mass index between 18.0 and 35 kg/m², both inclusive. Telephone Screen

Exclusion Criteria:

1. Currently undergoing medical treatment, including prescription drugs/medication. Medical History Interview
2. Clinically significant abnormal hematology, biochemistry, urinalysis, or coagulation screening tests, as judged by the Investigator. Medical History Interview
3. History or presence of cancer (except basal cell skin cancer or squamous cell skin cancer), or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological (with the exception euthyroid struma), haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders as judged by the Investigator. Medical History Interview
4. Seated blood pressure at screening (after resting for 5 min in seated position) outside the range of 90-140 mmHg for systolic or 50-90 mmHg for diastolic (excluding white-coat hypertension; therefore, if a repeated measurement shows values within the range, the subject can be included in the trial) and/or resting supine heart rate outside the range 50-90 beats per minute. Measurement taken at consent before eligibility is determined
5. Current Depression or Anxiety Symptoms using PHQ-8 (eight-item Patient Health Questionnaire depression scale) and GAD-7 (Generalized Anxiety Disorder 7-item scale). PHQ-8 score >= 10 and/or GAD-7 score >= 10 are excluded.

   (Past history of disorders not exclusionary). Interview
6. Currently taking SSRI (selective serotonin reuptake inhibitor) medications for any reason. Interview
7. Heart Diseases. Medical History Interview
8. Hepatitis B or C positive status. Medical History Interview
9. HIV positive status. Medical History Interview
10. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction. Medical History Interview
11. Use of non-prescription medication, herbal products or nutritional supplements during the study, and within the last 4 weeks before the start of the study (screening), as judged by the Investigator; occasional use of aspirin, ibuprofen, acetaminophen is permitted. Interview
12. Adherence to a vegan or vegetarian diet or to specialty/uncommon diets. Interview
13. Food Allergies to tree nuts, soy, cocoa and cocoa-containing products. Interview
14. People who choose to avoid caffeine intake. Interview
15. Current or history of alcoholism or drug/chemical abuse as per Investigator's judgment. Medical History Interview
16. Hormone Replacement Therapy; Currently pregnant; Pregnant or lactating within past 6 mos; Hormonal birth control (pill). Interview
17. Smoking. Interview
18. Unwilling to have blood drawn or anxiety/nausea during a blood draw. Interview.
19. Uncomfortable completing memory and attention tasks in the English language. Interview
20. MoCA (Montreal Cognitive Assessment) score less than 26. Montreal Cognitive Assessment
21. Inability to swallow study capsules. Interview (at consent).
22. Did not complete the two weeks Run-In Period (Participants who missed more than 2 intake occasions out of 14 days (28 occasions total) or if there are > 8 capsules left in the bottle after the two weeks will be excluded). Run-In Period.

MRI RELATED

1. Cardiac Pacemaker Interview
2. Internal Pump Interview
3. Insulin Pump Interview
4. Tattoo eyeliner Interview
5. Wire sutures Interview
6. Internal Metal Objects Interview
7. Metal Slivers in Eye Interview
8. Prosthesis Interview
9. Hearing Aid Implants Interview
10. Neurostimulator Interview
11. Metal Fragments Interview
12. Brain Aneurysm Clips Interview
13. Vascular Clips Interview
14. Breast Expander Interview
15. Vena Cava Filter Interview
16. Heart Valve Interview
17. Metal Stents Interview
18. Asthma Interview
19. Hay-Fever Interview
20. Sickle Cell Disease Interview
21. Kidney Disease Interview
22. Pregnant Interview
23. Claustrophobic Interview
24. Wheelchair bound Interview
25. Machinist or ever worked with heavy metals Interview
26. Contraindication to Gadolinium, including prior adverse reaction to gadolinium, past or current history of severe breathing difficulty that has been treated by a physician (e.g. asthma, COPD (Chronic obstructive pulmonary disease), etc) and sickle cell disease. History of renal impairment or estimated glomerular filtration rate <30 L/min.1.732m2 is also exclusionary Interview; Glomerular filtration rate assessed with creatinine via StatSensor monitor
27. Had more than one previous MRI scans with Gadolinium Interview

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Small, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Brickman AM, Khan UA, Provenzano FA, Yeung LK, Suzuki W, Schroeter H, Wall M, Sloan RP, Small SA. Enhancing dentate gyrus function with dietary flavanols improves cognition in older adults. Nat Neurosci. 2014 Dec;17(12):1798-803. doi: 10.1038/nn.3850. Epub 2014 Oct 26. PMID 25344629
- [Background] Bussy U , May BR , Olanrewaju Y , Hewitt G , Anderson N , Crozier A , Ottaviani JI , Kwik-Uribe C . Reliable, accessible and transferable method for the quantification of flavanols and procyanidins in foodstuffs and dietary supplements. Food Funct. 2020 Jan 29;11(1):131-138. doi: 10.1039/c9fo02762a. PMID 31932823
- [Background] Ottaviani JI, Fong R, Kimball J, Ensunsa JL, Britten A, Lucarelli D, Luben R, Grace PB, Mawson DH, Tym A, Wierzbicki A, Khaw KT, Schroeter H, Kuhnle GGC. Evaluation at scale of microbiome-derived metabolites as biomarker of flavan-3-ol intake in epidemiological studies. Sci Rep. 2018 Jun 29;8(1):9859. doi: 10.1038/s41598-018-28333-w. PMID 29959422

RESULTS

PARTICIPANT FLOW:
Recruitment Details: first consent; 1/13/2016 Final data collection session: 11/21/2018
  All data collected at Columbia University Medical Center
Pre-assignment Details: 1. consent: exclusions: 5 BMI too high; 66 MOCA too low; 4 elevated blood pressure; 16 other; 17 lost to follow-up
  2. two week run-in period: exclusions: 24 failed, 17 withdrew or lost to follow-up
  3. baseline assessments: exclusions: 1 lost to follow-up
Groups:
- 0 mg Cocoa Flavanol: daily consumption of capsules containing 0 mg cocoa flavanol for 12 weeks
- 260 mg Cocoa Flavanol: daily consumption of capsules containing 260 mg cocoa flavanol for 12 weeks;
- 510 mg Cocoa Flavanol: daily consumption of capsules containing 510 mg cocoa flavanol for 12 weeks;
- 770 mg Cocoa Flavanol: daily consumption of capsules containing 770 mg cocoa flavanol for 12 weeks;
Period: Overall Study
Arm/Group | 0 mg Cocoa Flavanol | 260 mg Cocoa Flavanol | 510 mg Cocoa Flavanol | 770 mg Cocoa Flavanol
Started | 53 | 53 | 53 | 52
Completed | 51 | 51 | 50 | 52
Not Completed | 2 | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- 0 mg: daily consumption of capsules containing 0 mg cocoa flavanol for 12 weeks
- 260 mg: daily consumption of capsules containing 260 mg cocoa flavanol for 12 weeks;
- 510 mg: daily consumption of capsules containing 510 mg cocoa flavanol for 12 weeks;
- 770 mg: daily consumption of capsules containing 770 mg cocoa flavanol for 12 weeks;
- Total: Total of all reporting groups
Arm/Group | 0 mg | 260 mg | 510 mg | 770 mg | Total
Number analyzed (Participants) | 53 | 53 | 53 | 52 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.47 (6.78) | 60.81 (6.71) | 61 (6.15) | 61.23 (6.37) | 61.13 (6.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 30 | 29 | 120
  Male | 22 | 23 | 23 | 23 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8 | 4 | 20
  Not Hispanic or Latino | 49 | 49 | 45 | 48 | 191
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 2 | 4 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 7 | 7 | 8 | 8 | 30
  White | 41 | 40 | 38 | 41 | 160
  More than one race | 1 | 3 | 3 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 53 | 53 | 52 | 211
alternative Healthy Eating Index (aHEI) [Mean (Standard Deviation); unit: units on a scale] — We used the Block 2005 food frequency questionnaire (FFQ) (NutritionQuest, Berkeley CA) to estimate customary dietary intake. The food list for this questionnaire was developed from the NHANES III dietary recall data. The nutrient database was developed from the USDA (United States Department of Agriculture) Nutrient Database for Standard Reference. Individual portion size was measured using pictures provided. From these data, we computed the alternative Healthy Eating Index (aHEI). The total aHEI score ranged from 0 (nonadherence) to 110 (perfect adherence).
  units on a scale | 65.09 (11.44) | 68.78 (10.82) | 64.83 (14.3) | 66.74 (10.84) | 66.36 (12)
5-(3',4'-dihydroxyphenyl)-γ-valerolactone (gVLM) [Mean (Standard Deviation); unit: nM] — gVLM is a nutritional biomarker of flavan-3-ol intake. Detection was achieved with a Waters Quattro Micromass spectrometer fitted with an electrospray interface (ESI; Waters). MS analysis was carried out in negative ionization mode by multiple reaction monitoring (MRM). Detection of gVL-3'-sulphate and -3'-O- glucuronide utilized transitions from 287 m/z to 207 m/z and 383 m/z to 207 m/z, respectively, and both with a dwell time of 0.02 s, a cone voltage of 32 V, and a collision energy of 20 V.
  nM | 19.7 (24.23) | 20.98 (34.28) | 44.32 (72.4) | 36.59 (72.06) | 30.44 (55.84)

OUTCOME MEASURES:

1. Primary Outcome: Modified Benton Recognition Task (ModBent)
Description: The ModBent task is divided into two parts. During the matching trials (top), participants were shown a complex stimulus for 10 s. Following a 1-s inter-trial interval, they were required to select, via a key press, which of two stimuli matched the one they had just studied, as quickly and as accurately as possible. Following 41 matching trials, participants were shown a series of 82 stimuli (bottom), 41 of which appeared on the initial study set during the matching trials and 41 of which were foils. They were required to indicate, as quickly as possible, whether each stimulus appeared earlier (yes response) or was new (no response). The primary variable of the ModBent task is the mean RT for correct rejections of foils during the recognition trials
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | 0 mg Cocoa Flavanol | 260 mg Cocoa Flavanol | 510 mg Cocoa Flavanol | 770 mg Cocoa Flavanol
Number analyzed (Participants) | 51 | 51 | 50 | 52
ms
  Baseline | 2807.98 (1733.36) | 2579.94 (1026.18) | 2603.65 (999.31) | 2732.79 (1367.96)
  12 Weeks | 2671.50 (1431.17) | 2489.84 (1135.40) | 2381.68 (929.14) | 2653.01 (1289.18)
Statistical Analysis 1: Comparison: 0 mg Cocoa Flavanol vs 260 mg Cocoa Flavanol vs 510 mg Cocoa Flavanol vs 770 mg Cocoa Flavanol; Test type: Superiority — Test of trend across doses; p = .393, Mixed Models Analysis; Change in outcome from baseline to 12 weeks tested using mixed effects models controlling for baseline measures, treatment, sex, age, and education; The flavanol effect on the change in each outcome from baseline to 12 weeks was tested using linear mixed effects models controlling for the respective baseline measures, four categories of treatment, sex, age, and education. Regression adjusted mean within-group tests of change were estimated and tested for statistical significance from the model. The primary test used for assessing the treatment effect was the linear trend contrast from the model across: placebo, low, medium and high dose. The model for cognitive measures incorporated additional outcome measurement times at 4 weeks and 20 weeks and included categorical time (4, 12, 20 weeks) as a predictor as well as a treatment (4 category) by time interaction, and a random intercept to control for repeated measures within individuals (results for 4 and 20 weeks not presented)

2. Secondary Outcome: Dentate Gyrus Cerebral Blood Volume
Description: measured in functional MRI. we generated high-resolution CBV brain maps using gadolinium-enhanced T1-weighted scans acquired perpendicular to the hippocampal long-axis, with sub-millimeter in-plane resolution of 0.68 × 0.68 mm and slice thickness of 3 mm. To perform group-wise voxel-based analyses on the whole hippocampal circuit, we first isolated hippocampal subfields using FreeSurfer segmentations and thresholded posterior probabilities to generate a composite mask of the bilateral hippocampal formation. These masked T1-weighted images were then used to generate a group-wise template to which individual images were co-registered using a diffeomorphic technique that maximizes cross-correlation among images.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: % cerebral blood volume
Arm/Group | 0 mg Cocoa Flavanol | 260 mg Cocoa Flavanol | 510 mg Cocoa Flavanol | 770 mg Cocoa Flavanol
Number analyzed (Participants) | 14 | 10 | 13 | 12
% cerebral blood volume
  Baseline | 2.44 (.81) | 2.17 (.69) | 2.11 (0.47) | 1.85 (0.67)
  12 Weeks | 2.25 (.57) | 2.11 (.52) | 2.01 (.71) | 2.23 (.59)

3. Secondary Outcome: Modified Benton Recognition Task (ModBent)
Description: as for outcome 1
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | 0 mg Cocoa Flavanol | 260 mg Cocoa Flavanol | 510 mg Cocoa Flavanol | 770 mg Cocoa Flavanol
Number analyzed (Participants) | 50 | 49 | 50 | 51
ms | 2542.76 (1278.87) | 2475.35 (1512.88) | 2373.78 (934.84) | 2550.18 (1165.92)

4. Secondary Outcome: Modified Rey Auditory Verbal Learning Test
Description: In learning Trials 1 to 3 the participant is read 20 unique, semantically/phonemically unrelated words (List A) and is to free recall those words after each trial. Next the participant is read a list of 20 unique words (List B) and is to recall as many as possible. This trial is followed by a short delay free recall trial: the participant is to recall as many words as possible from List A. After a 1.5-hour, the participant is asked to long delay free recall words from List A and then from List B. This is followed by a 66-item forced recognition trial: the participant is read a list of 66 words and asked to distinguish List A words from semantic and phonemic distractors, including words from List B. Finally, a source memory trial is administered: the examiner serially reads words from List A and B. The participant is to specify from which list each word came.Higher score indicates better performance. score ranges from 0 to 60.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0 mg | 260 mg | 510 mg | 770 mg
Number analyzed (Participants) | 51 | 51 | 50 | 52
units on a scale
  Baseline | 38.91 (8.45) | 37.25 (8.19) | 39.75 (7.38) | 39.96 (9.62)
  12 Weeks | 39.49 (9.70) | 38.69 (9.30) | 41.10 (8.50) | 41.92 (8.48)

5. Secondary Outcome: NIH Toolbox Cognition Battery (NIHTB-CB): The List Sorting Test
Description: Participants are presented with a series of stimuli, each of which is both visually and auditorily presented by computer. A picture of each stimulus is displayed on the computer monitor for 2 seconds while the name of the stimulus is simultaneously being read via a computerized voice; stimuli are presented one after another. The participant must remember each stimulus in a series, mentally reorder them from smallest to largest, and recite the names of the stimuli in this order. List Sorting scores are based upon Total Score. Higher score indicated better performance.Score ranges from 0-100.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0 mg | 260 mg | 510 mg | 770 mg
Number analyzed (Participants) | 51 | 51 | 50 | 52
units on a scale
  Baseline | 52.89 (8.85) | 56.81 (8.91) | 54.60 (9.15) | 55.18 (8.65)
  12 Weeks | 53.34 (7.44) | 56.10 (8.47) | 54.86 (8.56) | 53.46 (9.23)

ADVERSE EVENTS:
Time Frame: adverse events were monitored each week throughout the study and for the MRI substudy, at each of the two MRI sessions
Arm/Group | 0 mg Cocoa Flavanol | 260 mg Cocoa Flavanol | 510 mg Cocoa Flavanol | 770 mg Cocoa Flavanol
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53 | 0/53 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53 | 0/53 | 0/52
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53 | 0/53 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT02312310/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT02312310/SAP_001.pdf